CLINICAL TRIAL: NCT06472817
Title: iCCARE Project # 4: Grounded Theory Study of the Social Determinants of Migrant Health Factors Impacting Prostate Cancer Care and Survivorship Among Sub-Saharan African and Caribbean Immigrant Men Diagnosed With Prostate Cancer
Brief Title: Social Determinants of Migrant Health Factors Impacting Prostate Cancer Care and Survivorship Among Sub-Saharan African and Caribbean Immigrant Men
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 22-005329; NCI-2024-03996 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17109 (Other: Mayo Clinic); 22-005329 (Other: Mayo Clinic Institutional Review Board); W81XWH-22-1-0971 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: AIM I: Participants complete a survey and participate in an interview in person, over the phone, or via zoom on study.
  AIM II: Participants complete an interview in person, over the phone, or via zoom on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study is being done to understand what social factors affect health decisions for those who have immigrated from another country by examining how the immigration from Sub-Sahara Africa affects the experiences of participants regarding health-seeking behaviors, care, and treatment of prostate cancer. It also examines similarities and differences among participants based on their region of origin in Africa.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To employ the social determinant of migrant health framework (International Organization for Migration, n.d.) to examine the impact of immigration on the health-seeking behaviors of SSAI including informed-decision making, psychosocial effects and coping mechanisms. (Phase I) II. To examine SDOMH factors among SSAI and CI men, including their migration experience and health behaviors. (Phase II)

OUTLINE: This is an observational study.

AIM I: Participants complete a survey and participate in an interview in person, over the phone, or via zoom on study.

AIM II: Participants complete an interview in person, over the phone, or via zoom on study.

ELIGIBILITY:
Inclusion Criteria:

* PHASE I:

  * Adult men originally from each of these geographic regions (East, West, Central, and Southern Africa) and have been diagnosed with prostate cancer
  * Able to provide written consent and conduct an interview
  * Able to speak and understand English
* PHASE II:

  * Caribbean Immigrant men and SSAI men diagnosed with CaP within the last 10 years who identify as Black and speak English
  * Able to provide written consent and conduct an interview
  * Able to speak and understand English

Exclusion Criteria:

* PHASE I:

  * Patients below the ages of 18, and those not belonging to any of four regions
  * Employees of Mayo Clinic will be excluded
  * Non-English speakers will not be included
* PHASE II:

  * Individuals below the age of 18
  * Those not diagnosed with prostate cancer and individuals not from the regions described above
  * Employees of Mayo Clinic will be excluded
  * Non-English speakers will not be included

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sub-Saharan African immigrant men who were diagnosed with prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2026-09-11 (Estimated); Study Completion 2026-09-11 (Estimated)

PRIMARY OUTCOMES:
Qualitative Interview - identification of themes and constructs | Baseline
  Data will be collected during an in-depth interview and will be analyzed with an inductive, open coding approach, first identifying themes, then constructs that emerge from the data will be categorized and mapped, noting new concepts and constructs. Theme convergence and divergence will be assessed. The interview guide focuses on participants' experiences and health-seeking behaviors regarding prostate cancer prevention, detection, decision-making, treatment, care, and survivorship.
Immigrant social determinants of health factors that impact Sub-Saharan African Immigrant (SSAI) carcinoma of the prostate (CaP) survivors | Baseline
  From the data generated in Outcome 1 interviews, an interpretive framework or theoretical model for SSAI men will be developed to evaluate and identify factors that contribute to or exacerbate disparities in prostate cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Gladys B. Asiedu, Ph.D., Principal Investigator — Mayo Clinic in Rochester
Locations (2):
- United States (2):
  - Georgia State University, Atlanta, Georgia
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials